CLINICAL TRIAL: NCT00877526
Title: DiabCare Asia 2008 (Malaysia): A Cross-Sectional Survey to Evaluate Diabetes Management, Control, Complications, Psychosocial Aspects of Diabetic Patients in Asia & To Evaluate Perceptions and Practices of Physicians & Patients About Diabetes Management in Asia
Brief Title: A Survey to Evaluate Diabetes Management, Control, Chronic Complications, Psychosocial Aspects of Diabetic Subjects in Malaysia
Acronym: DiabCare Asia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3723
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Capillary or venous blood will be drawn for analysing HbA1c.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Subject will only fill out a questionaire when entering the observational study.

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate current status of diabetes management, control, and complications in diabetic subjects in Asia.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients registered in the particular centre for more than 12 months.
* Patients should have visited the centre at least once in the last 3-6 months apart from the initial visit.
* Patients willing to sign informed consent form.

Exclusion Criteria:

* Repetition of any patient as patients should not be included twice for any reason.
* Unwilling to participate or unable to comply with protocol requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus (both type 1 and type 2) being treated at general hospitals, diabetes clinics and referral clinics will be selected according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1670 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Mean age of onset of type 1 and type 2 diabetes mellitus, respectively | at baseline visit/study start
Mean duration of treatment of type 2 Diabetes mellitus | at baseline visit/study start
Percentage of patients on insulin and Oral Anti-Diabetics Drugs (OADs) theraphy, respectively | at baseline visit/study start
Mean duration of diabetes in type 1 and type 2 diabetic patients respectively | at baseline visit/study start
Mean FPG (Fasting plasma glucose), PPG (Post prandial glucose) and HbA1c of diabetic patients | at baseline visit/study start
Percentage of diabetic patients with HbA1c target below 7.0% and below 6.5%, respectively | at baseline visit/study start
Percentage of diabetic patients having dyslipidemia and hypertension, cardiovascular complications, peripheral vascular disease, diabetic nephropathy and diabetic eye complications, respectively | at baseline visit/study start

SECONDARY OUTCOMES:
Patients' perception will be analysed through patient questionnaire measuring: Psychological well-being, Quality of Life and patients' compliant to treatmen | at baseline visit/study start
Physician perception of diabetes and its management will be analysed through physician questionnaire measuring awareness about: HbA1c test and its goal, anti-diabetic treatment, barriers towards optimum diabetes control | at baseline visit/study start
Duration of diabetes associated with highest number of diabetic complications | at baseline visit/study start
Minimum duration of diabetes associated with 10% incidence of diabetic complications (CVD, Nephropathy and retinopathy) | at baseline visit/study start

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Selangor Darul Ehsan, Malaysia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com